CLINICAL TRIAL: NCT01143051
Title: Phase I/II Study Epinephrine Inhalation Aerosol USP, an HFA-MDI Clinical Study-B for Assessment of Pharmacokinetics
Brief Title: Pharmacokinetics (PK) Study of Epinephrine Inhalation Aerosol in Healthy Volunteers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amphastar Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: API-E004-CL-B
Record Dates: First submitted 2010-06-07; First posted 2010-06-14 (Estimated); Results first posted 2014-07-15 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Asthma
Keywords: Asthma; Pharmacokinetics; Epinephrine; Bronchodilator; metered dose inhaler
MeSH Terms: conditions — Asthma | interventions — Epinephrine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment C (Active Comparator): Active comparator arm utilizing marketed Primatene Mist with CFC propellant at the labeled dose.
  Interventions: Drug: epinephrine inhalation aerosol
- Treatment 1 (Experimental): T1 is HFA propelled epinephrine inhalation aerosol 125 mcg/inhalation
  Interventions: Drug: epinephrine inhalation aerosol
- Treatment 2 (Experimental): HFA propelled epinephrine inhalation aerosol, 160 mcg/inhalation
  Interventions: Drug: epinephrine inhalation aerosol

INTERVENTIONS:
Drug: epinephrine inhalation aerosol — Single dose 220 mcg/inhalation, 10 inhalations
  Other Names: Primatene Mist
  Arms: Treatment C
Drug: epinephrine inhalation aerosol — HFA propelled epinephrine inhalation aerosol, 125 mcg/inhalation, 10 inhalations
  Other Names: Primatene Mist
  Arms: Treatment 1
Drug: epinephrine inhalation aerosol — HFA propelled epinephrine inhalation aerosol, 160 mcg/inhalation, 10 inhalations
  Other Names: Primatene Mist
  Arms: Treatment 2

SUMMARY:
This study examines the pharmacokinetic profile of Armstrong's proposed Epinephrine Inhalation Aerosol USP, an HFA-MDI (E004), in healthy male and female adult volunteers. Safety of E004 will also be evaluated, under augmented dose conditions.

DETAILED DESCRIPTION:
This study is a randomized, evaluator-blind, single dose, three-arm, crossover, PK study, to be conducted in ~18 healthy, male and female, adult volunteers. PK will be studied at two dose strengths (Arm T1 and Arm T2). A currently marketed, non-labeled, Epinephrine CFC-MDI will be used as a Reference Control (Arm C).

* At the Screening Visit and the beginning of each Study Visit, each subject will be trained on the correct self-administration of MDI. The following three randomized treatments will be self-administered, at three Study Visits:

  * Treatment T1: Ten (10) inhalations of the low dose E004(125 mcg/inhalation), totaling 1.25 mg of epinephrine;
  * Treatment T2: Ten (10) inhalations of the high dose E004 (160 mcg/inhalation), totaling 1.60 mg of epinephrine;
  * Treatment C: Ten (10) inhalations of Epinephrine CFC-MDI (220 mcg/inhalation, totaling 2.2 mg of epinephrine base equivalent).
* PK blood samples will be taken from a vein at scheduled time points.
* Safety parameters and adverse drug events, if any, will be monitored and documented at each study visit. An End-of-Study (EOS) safety evaluation will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy, male and female adults, 18-30 yrs of age at Screening;
* Having no clinically significant respiratory, cardiovascular and other systemic or organic illnesses, per investigator discretion;
* Women of child-bearing potential must be non-pregnant, non-lactating, and practicing a clinically acceptable form of birth control;
* Having properly consented and satisfied all other inclusion/exclusion criteria as required for this protocol.
* Other criteria apply.

Exclusion Criteria:

* A recent or significant smoking history;
* Use of prohibited drugs or failure to observe the drug washout restrictions;
* Having been on other investigational drug/device studies in the last 30 days prior to Screening.
* Other criteria apply

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Amphastar Pharmaceuticals, Inc.
Locations (1):
- Amphastar Location 1, Cypress, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from a specialty clinic in Cypress, CA between 04/29/2010 and 05/27/2010
Pre-assignment Details: A total of 38 subjects were screened, 24 subjects passed screening, consented and were randomized for participation in the study. The IRB approval date was 04/29/2010, the last subject was screened on 05/27/2010.
Groups:
- C, T1, T2: Subjects received one of the three treatments during each study visit, separated by a washout period of 3-14 days. Visit 1: Treatment C: Ten (10) inhalations of Epinephrine CFC-MDI (220 mcg/inhalation), totaling 2.20 mg of epinephrine, in 5 min; Visit 2: Treatment T1: Ten (10) inhalations of the low dose E004 (125 mcg/inhalation), totaling 1.25 mg of epinephrine, in 5 min; Visit 3: Treatment T2: Ten (10) inhalations of the high dose E004 (160 mcg/inhalation), totaling 1.60 mg of epinephrine, in 5 min.
- C, T2, T1: Subjects received one of the three treatments during each study visit, separated by a washout period of 3-14 days. Visit 1: Treatment C: Ten (10) inhalations of Epinephrine CFC-MDI (220 mcg/inhalation), totaling 2.20 mg of epinephrine, in 5 min; Visit 2: Treatment T2: Ten (10) inhalations of the high dose E004 (160 mcg/inhalation), totaling 1.60 mg of epinephrine, in 5 min; Visit 3: Treatment T1: Ten (10) inhalations of the low dose E004 (125 mcg/inhalation), totaling 1.25 mg of epinephrine, in 5 min.
- T1, C, T2: Subjects received one of the three treatments during each study visit, separated by a washout period of 3-14 days. Visit 1: Treatment T1: Ten (10) inhalations of the low dose E004 (125 mcg/inhalation), totaling 1.25 mg of epinephrine, in 5 min; Visit 2: Treatment C: Ten (10) inhalations of Epinephrine CFC-MDI (220 mcg/inhalation), totaling 2.20 mg of epinephrine, in 5 min; Visit 3: Treatment T2: Ten (10) inhalations of the high dose E004 (160 mcg/inhalation), totaling 1.60 mg of epinephrine, in 5 min.
- T1, T2, C: Subjects received one of the three treatments during each study visit, separated by a washout period of 3-14 days. Visit 1: Treatment T1: Ten (10) inhalations of the low dose E004 (125 mcg/inhalation), totaling 1.25 mg of epinephrine, in 5 min; Visit 2: Treatment T2: Ten (10) inhalations of the high dose E004 (160 mcg/inhalation), totaling 1.60 mg of epinephrine, in 5 min; Visit 3: Treatment C: Ten (10) inhalations of Epinephrine CFC-MDI (220 mcg/inhalation), totaling 2.20 mg of epinephrine, in 5 min.
- T2, C, T1: Subjects received one of the three treatments during each study visit, separated by a washout period of 3-14 days. Visit 1: Treatment T2: Ten (10) inhalations of the high dose E004 (160 mcg/inhalation), totaling 1.60 mg of epinephrine, in 5 min; Visit 2: Treatment C: Ten (10) inhalations of Epinephrine CFC-MDI (220 mcg/inhalation), totaling 2.20 mg of epinephrine, in 5 min; Visit 3: Treatment T1: Ten (10) inhalations of the low dose E004 (125 mcg/inhalation), totaling 1.25 mg of epinephrine, in 5 min.
- T2, T1, C: Subjects received one of the three treatments during each study visit, separated by a washout period of 3-14 days. Visit 1: Treatment T2: Ten (10) inhalations of the high dose E004 (160 mcg/inhalation), totaling 1.60 mg of epinephrine, in 5 min; Visit 2: Treatment T1: Ten (10) inhalations of the low dose E004 (125 mcg/inhalation), totaling 1.25 mg of epinephrine, in 5 min; Visit 3 Treatment C: Ten (10) inhalations of Epinephrine CFC-MDI (220 mcg/inhalation), totaling 2.20 mg of epinephrine, in 5 min.
Period: Visit 1
Arm/Group | C, T1, T2 | C, T2, T1 | T1, C, T2 | T1, T2, C | T2, C, T1 | T2, T1, C
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: 3-14 Day Washout
Arm/Group | C, T1, T2 | C, T2, T1 | T1, C, T2 | T1, T2, C | T2, C, T1 | T2, T1, C
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 3 | 4 | 4 | 4
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0
Period: Visit 2
Arm/Group | C, T1, T2 | C, T2, T1 | T1, C, T2 | T1, T2, C | T2, C, T1 | T2, T1, C
Started | 4 | 4 | 3 | 4 | 4 | 4
Completed | 4 | 4 | 3 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: 3-14 Day Washout
Arm/Group | C, T1, T2 | C, T2, T1 | T1, C, T2 | T1, T2, C | T2, C, T1 | T2, T1, C
Started | 4 | 4 | 3 | 4 | 4 | 4
Completed | 4 | 4 | 3 | 4 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1
Period: Visit 3
Arm/Group | C, T1, T2 | C, T2, T1 | T1, C, T2 | T1, T2, C | T2, C, T1 | T2, T1, C
Started | 4 | 4 | 3 | 4 | 4 | 3
Completed | 4 | 4 | 3 | 4 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | C, T1, T2 | C, T2, T1 | T1, C, T2 | T1, T2, C | T2, C, T1 | T2, T1, C | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 4 | 4 | 4 | 4 | 24
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.0 (2.94) | 25.3 (4.27) | 24.0 (3.37) | 21.8 (1.71) | 25.3 (0.50) | 22.0 (3.56) | 23.7 (3.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 2 | 1 | 2 | 9
  Male | 3 | 2 | 3 | 2 | 3 | 2 | 15
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 4 | 4 | 4 | 4 | 24

OUTCOME MEASURES:

1. Primary Outcome: Baseline Concentration (C0) of Labeled Epinephrine Total Epinephrine
Description: Patient PK blood samples were taken from a vein in a hand or arm via indwelling heparin-anticoagulated IV catheters, or by venipunctures at Baseline (prior to dosing) in each treatment period following a specified washout period (3-14 days), and were analyzed using an established analysis method. Baseline concentration (C0) is the concentration of epinephrine measured in the plasma at this time point.
Time Frame: 0 to 30 minutes prior to dosing
Population: Patients who: 1) have taken the valid pre-dose baseline PK sample 2) have correctly taken the randomized study-drug treatment 3) have at least four of the five post-dose PK measurements between 5 and 60 min post-dose available and 4) have a minimum of eight of the ten post-dose PK measurements for the entire 6 hour post-dose PK sampling period.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Treatment T1: Ten (10) inhalations of the low dose E004 (125 mcg/inhalation), totaling 1.25 mg of epinephrine
- Treatment T2: Ten (10) inhalations of the high dose E004 (160 mcg/inhalation), totaling 1.60 mg of epinephrine
- Treatment C: Ten(10) inhalations of Epinephrine CFC-MDI (220 mcg/inhalation), totaling 2.20 mg of epinephrine
Arm/Group | Treatment T1 | Treatment T2 | Treatment C
Number analyzed (Participants) | 24 | 22 | 22
pg/mL | 9.3 (17.7) | 8.9 (15.8) | 7.8 (21.4)

2. Primary Outcome: Area Under the Curve From Time Zero to 6 Hours Post-dose (AUC[0-6])
Description: Patient PK blood samples were taken from a vein in a hand or arm via indwelling heparin-anticoagulated IV catheters, or by venipunctures at 0 (baseline), 5, 15, 30, 45, 60, 90, 120, 180, 240, and 360 minutes post-dose in each treatment period and were analyzed using an established analysis method. Area under the curve from time zero to 6 hours post-dose (AUC[0-6]) was calculated using the trapezoidal rule.
Time Frame: Pre-dose to 6 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg*min/mL
Arm/Group | Treatment T1 | Treatment T2 | Treatment C
Number analyzed (Participants) | 24 | 22 | 22
pg*min/mL | 7938 (5023) | 9438 (4819) | 7218 (6489)

3. Primary Outcome: Peak Concentration (Cmax) for Total Epinephrine From Time Zero to 6 Hours Post-dose
Description: Patient PK blood samples were taken from a vein in a hand or arm via indwelling heparin-anticoagulated IV catheters, or by venipunctures at 0 (baseline), 5, 15, 30, 45, 60, 90, 120, 180, 240, and 360 minutes post-dose in each treatment period and were analyzed using an established analysis method. Peak (maximum) concentration (Cmax) is the highest concentration of epinephrine measured in plasma during the treatment period.
Time Frame: Pre-dose to 6 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Treatment T1 | Treatment T2 | Treatment C
Number analyzed (Participants) | 24 | 22 | 22
pg/mL | 340 (294) | 444 (328) | 139 (98)

4. Primary Outcome: Time to Reach Peak Concentration (Tmax) for Total Epinephrine
Description: Patient PK blood samples were taken from a vein in a hand or arm via indwelling heparin-anticoagulated IV catheters, or by venipunctures at 0 (baseline), 5, 15, 30, 45, 60, 90, 120, 180, 240, and 360 minutes post-dose in each treatment period and were analyzed using an established analysis method. tmax is the amount of time it takes for epinephrine to reach peak concentration in plasma during the treatment period.
Time Frame: Pre-dose to 6 hours post-dose
Population: Patients who : 1) have taken the valid pre-dose baseline PK sample 2) have correctly taken the randomized study-drug treatment 3) have at least four of the five post-dose PK measurements between 5 and 60 min post-dose available and 4) have a minimum of eight of the ten post-dose PK measurements for the entire 6 hour post-dose PK sampling period.
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Treatment T1 | Treatment T2 | Treatment C
Number analyzed (Participants) | 24 | 22 | 22
min | 34.6 (100.2) | 37.0 (104.5) | 38.0 (104.3)

5. Primary Outcome: Half-life (t1/2) for Total Epinephrine
Description: Patient PK blood samples were taken from a vein in a hand or arm via indwelling heparin-anticoagulated IV catheters, or by venipunctures at 0 (baseline), 5, 15, 30, 45, 60, 90, 120, 180, 240, and 360 minutes post-dose in each treatment period and were analyzed using an established analysis method. Half-life (t1/2) is the amount of time it takes for epinephrine decrease to half the peak concentration in plasma during the treatment period.
Time Frame: Pre-dose to 6 hours post-dose
Population: Patients who: 1) have taken the valid pre-dose baseline PK sample 2) have correctly taken the randomized study-drug treatment 3) have at least 4 of the 5 post-dose PK measurements between 5 and 60 min post-dose available; and 4) have a min of 8 of the 10 post-dose PK measurements for the entire 6 hour post-dose PK sampling period.
Measure: Mean (Full Range); unit: min
Arm/Group | Treatment T1 | Treatment T2 | Treatment C
Number analyzed (Participants) | 24 | 22 | 22
min | 125.9 (183.3) [10.8 to 337.3] | 158.8 (238.0) [3.1 to 432.8] | 237.3 (175.2) [6.8 to 490.2]

6. Primary Outcome: Concentration vs. Time for Total Epinephrine From Time Zero to 6 Hours Post-dose
Description: Patient PK blood samples were taken from a vein in a hand or arm via indwelling heparin-anticoagulated IV catheters, or by venipunctures at 0 (baseline), 5, 15, 30, 45, 60, 90, 120, 180, 240, and 360 minutes post-dose in each treatment period and were analyzed using an established analysis method.
Time Frame: Pre-dose to 6 hours post-dose
Population: Patients who : 1) have taken the valid pre-dose baseline PK sample 2) have correctly taken the randomized study-drug treatment 3) have at least 4 of the 5 post-dose PK measurements between 5 and 60 minutes post-dose available and 4) have a min of 8 of the 10 post-dose PK measurements for the entire 6 hour post-dose PK sampling period.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Treatment T1 | Treatment T2 | Treatment C
Number analyzed (Participants) | 24 | 22 | 22
pg/mL
  Total Epinephrine, 0 min (Baseline) | 9.3 (17.7) | 8.9 (15.8) | 7.8 (21.4)
  Total Epinephrine, 5 min post-dose | 339.6 (295.1) | 442.4 (330.8) | 130.2 (101.8)
  Total Epinephrine, 15 min post-dose | 48.9 (33.7) | 62.4 (42.5) | 38.5 (21.2)
  Total Epinephrine, 30 min post-dose | 12.7 (18.8) | 17.4 (18.3) | 16.8 (17.6)
  Total Epinephrine, 45 min post-dose | 8.6 (14.4) | 13.0 (17.2) | 20.9 (18.6)
  Total Epinephrine, 60 min post-dose | 7.6 (14.7) | 14.5 (17.3) | 18.0 (18.6)
  Total Epinephrine, 90 min post-dose | 5.7 (11.6) | 13.7 (14.8) | 16.7 (16.6)
  Total Epinephrine, 120 min post-dose | 8.7 (12.8) | 15.5 (19.7) | 13.1 (17.6)
  Total Epinephrine, 180 min post-dose | 12.0 (20.2) | 10.4 (15.2) | 8.4 (15.2)
  Total Epinephrine, 240 min post-dose | 12.9 (20.4) | 11.5 (14.9) | 9.8 (18.1)
  Total Epinephrine, 360 min post-dose | 31.1 (24.0) | 29.4 (23.0) | 38.3 (40.8)

7. Secondary Outcome: Vital Signs: Systolic Blood Pressure (SBP)
Description: Subject vital signs, i.e., blood pressure and heart rate, were measured prior to study drug dosing (baseline) and up to 360 minutes after dosing during the study visit.
Time Frame: Pre-dose (baseline) to 360 minutes post-dose
Population: Subjects who have taken any amount of study drug treatment.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Treatment C: Ten (10) inhalations of Epinephrine CFC-MDI (220 mcg/inhalation), totaling 2.20 mg of epinephrine
Arm/Group | Treatment T1 | Treatment T2 | Treatment C
Number analyzed (Participants) | 24 | 23 | 22
mmHg
  Pre-dose (Baseline) | 110 (10.0) | 112 (13.2) | 111 (9.4)
  10 min post-dose | 123 (13.8) | 122 (14.1) | 121 (11.3)
  30 min post-dose | 116 (12.3) | 117 (11.5) | 116 (10.6)
  60 min post-dose | 113 (11.2) | 113 (9.9) | 115 (10.0)
  120 min post-dose | 112 (10.4) | 114 (9.6) | 114 (10.9)
  180 min post-dose | 114 (10.1) | 113 (11.4) | 115 (11.0)
  360 min post-dose | 113 (9.8) | 113 (9.3) | 113 (9.5)

8. Secondary Outcome: Vital Signs: Diastolic Blood Pressure (DBP)
Description: as for outcome 7
Time Frame: Pre-dose (baseline) to 360 minutes post-dose
Population: Subjects who have taken any amount of study drug treatment.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Treatment T1 | Treatment T2 | Treatment C
Number analyzed (Participants) | 24 | 23 | 22
mmHg
  Pre-dose (Baseline) | 62 (9.3) | 61 (11.2) | 61 (10.8)
  10 min post-dose | 63 (10.1) | 64 (10.0) | 65 (10.2)
  30 min post-dose | 64 (11.2) | 64 (9.2) | 65 (9.5)
  60 min post-dose | 63 (10.8) | 64 (10.4) | 63 (8.8)
  120 min post-dose | 61 (9.8) | 63 (11.9) | 62 (10.6)
  180 min post-dose | 62 (8.3) | 60 (9.5) | 59 (7.5)
  360 min post-dose | 62 (8.8) | 62 (10.1) | 62 (8.0)

9. Secondary Outcome: Vital Signs: Heart Rate (HR)
Description: as for outcome 7
Time Frame: Pre-dose (baseline) to 360 minutes post-dose
Population: Subjects who have taken any amount of study drug treatment.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Treatment T1 | Treatment T2 | Treatment C
Number analyzed (Participants) | 24 | 23 | 22
beats per minute
  Pre-dose (Baseline) | 60 (10.1) | 62 (12.2) | 58 (11.7)
  10 min post-dose | 67 (14.0) | 69 (12.2) | 62 (12.7)
  30 min post-dose | 63 (14.2) | 64 (9.8) | 61 (13.7)
  60 min post-dose | 67 (12.9) | 67 (14.4) | 61 (10.8)
  120 min post-dose | 60 (10.1) | 60 (7.1) | 58 (9.4)
  180 min post-dose | 66 (11.1) | 66 (10.5) | 63 (9.9)
  360 min post-dose | 64 (8.7) | 64 (10.4) | 61 (8.4)

10. Secondary Outcome: ECG: QT Interval
Description: Subject QT and QTc Intervals were recorded using a 12-Lead ECG prior to study drug dosing (baseline) and up to 360 minutes after dosing during the study visit.
Time Frame: Pre-dose (baseline) to 360 minutes post-dose
Population: Subjects who have taken any amount of study drug treatment.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Treatment T1 | Treatment T2 | Treatment C
Number analyzed (Participants) | 24 | 23 | 22
msec
  Pre-dose (Baseline) | 416 (33.6) | 407 (30.1) | 423 (44.1)
  30 min post-dose | 404 (38.6) | 405 (32.8) | 413 (44.8)
  90 min post-dose | 399 (34.3) | 401 (32.9) | 407 (41.3)
  360 min post-dose | 399 (41.5) | 400 (33.1) | 400 (37.7)

11. Secondary Outcome: ECG: QTc Interval
Description: as for outcome 10
Time Frame: Pre-dose (baseline) to 360 minutes post-dose
Population: Subjects who have taken any amount of study drug treatment.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Treatment T1 | Treatment T2 | Treatment C
Number analyzed (Participants) | 24 | 23 | 22
msec
  Pre-dose (Baseline) | 407 (16.9) | 407 (20.0) | 403 (16.2)
  30 min post-dose | 408 (15.2) | 411 (19.4) | 412 (22.3)
  90 min post-dose | 401 (16.9) | 401 (18.1) | 403 (14.1)
  360 min post-dose | 403 (18.2) | 403 (17.9) | 402 (15.7)

12. Secondary Outcome: Serum Glucose Levels
Description: Blood samples used to measure subject serum glucose and potassium levels were collected prior to study drug dosing (baseline) and up to 360 minutes post-dose.
Time Frame: Pre-dose (baseline) to 360 minutes post-dose
Population: Subjects who have taken any amount of study drug treatment.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment T1 | Treatment T2 | Treatment C
Number analyzed (Participants) | 24 | 23 | 22
mg/dL
  Pre-dose (Baseline) | 83 (6.9) | 83 (9.1) | 84 (6.2)
  15 min post-dose | 101 (17.0) | 105 (11.6) | 96 (11.0)
  30 min post-dose | 94 (16.4) | 99 (12.1) | 98 (10.7)
  60 min post-dose | 86 (8.9) | 86 (10.8) | 94 (12.5)
  120 min post-dose | 81 (6.8) | 82 (6.1) | 83 (5.3)
  360 min post-dose | 82 (7.9) | 82 (9.4) | 80 (7.1)

13. Secondary Outcome: Serum Potassium Levels
Description: as for outcome 12
Time Frame: Pre-dose (baseline) to 360 minutes post-dose
Population: Subjects who have taken any amount of study drug treatment.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Treatment T1 | Treatment T2 | Treatment C
Number analyzed (Participants) | 24 | 23 | 22
mmol/L
  Pre-dose (Baseline) | 4 (0.2) | 4 (0.3) | 4 (0.2)
  15 min post-dose | 4 (0.3) | 4 (0.3) | 4 (0.3)
  30 min post-dose | 4 (0.5) | 4 (0.3) | 4 (0.3)
  60 min post-dose | 4 (0.2) | 4 (0.3) | 4 (0.2)
  120 min post-dose | 4 (0.3) | 4 (0.3) | 4 (0.3)
  360 min post-dose | 4 (0.3) | 4 (0.3) | 4 (0.2)

14. Secondary Outcome: Hand Tremor Scores
Description: Subjects evaluated hand tremor experiences using a scale from 0 to 3 (0: No tremor; 1: Mild, perceivable; 2: Moderate, observable; and 3: Severe, interfering with hand activities). Hand tremors were evaluated prior to study drug dosing (baseline) and up to 360 minutes post-dose.
Time Frame: Pre-dose (baseline) to 360 minutes post-dose
Population: Subjects who have taken any amount of study drug treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment T1 | Treatment T2 | Treatment C
Number analyzed (Participants) | 24 | 23 | 22
score on a scale
  Pre-dose (Baseline) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  10 min post-dose | 0.1 (0.3) | 0.2 (0.4) | 0.1 (0.4)
  60 min post-dose | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.2)
  360 min post-dose | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.2)

15. Secondary Outcome: Number of Subjects With Significant Changes in Physical Examination
Description: Physical examinations were performed as a part of Screening and End-of-Study (EOS) procedures. This outcome is a count of the number of subjects that showed a clinically significant change in the EOS physical examination compared to the Screening Visit.
Time Frame: Approximately 6 weeks
Population: Subjects who have taken any amount of study drug treatment. The Arm/Group is presented as one group because subjects would have received all 3 different study drug treatments prior to EOS due to the crossover study design.
Measure: Count of Participants; unit: Participants
Groups:
- Randomized Subjects: Subjects who have taken any amount of study drug treatment.
Arm/Group | Randomized Subjects
Number analyzed (Participants) | 24
Participants | 0

16. Secondary Outcome: Number of Subjects With Significant Changes in Laboratory Tests
Description: Laboratory tests (CBC, serum comprehensive metabolic panel, urinalysis, and urinary pregnancy test for women of childbearing potential) were performed as a part of Screening and End-of-Study (EOS) procedures. This outcome is a count of the number of subjects that showed a clinically significant change in the EOS laboratory tests compared to the Screening Visit.
Time Frame: Approximately 6 weeks
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Subjects
Number analyzed (Participants) | 24
Participants | 0

ADVERSE EVENTS:
Time Frame: All patients were closely monitored for any incidence of adverse events by the investigators during the entire study period.
Groups:
- Treatment T1: T1 is HFA propelled epinephrine inhalation aerosol 125 mcg/inhalation
  epinephrine inhalation aerosol : HFA propelled epinephrine inhalation aerosol, 125 mcg/inhalation, 10 inhalations
- Treatment T2: HFA propelled epinephrine inhalation aerosol, 160 mcg/inhalation
  epinephrine inhalation aerosol : HFA propelled epinephrine inhalation aerosol, 160 mcg/inhalation, 10 inhalations
- Treatment C: Active comparator arm utilizing marketed Primatene Mist with CFC propellant at the labeled dose.
  epinephrine inhalation aerosol : Single dose 220 mcg/inhalation, 10 inhalations
Arm/Group | Treatment T1 | Treatment T2 | Treatment C
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/23 | 0/22
Other Adverse Events (participants affected / at risk) | 1/24 | 1/23 | 1/22
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment T1 (N=24) | Treatment T2 (N=23) | Treatment C (N=22)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upset stomach (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sore throat (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lightheadedness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI is to maintain all information, data, inventions and discoveries disclosed by the Sponsor in confidence unless that information was in public domain at time of disclosure or becomes part of the public domain or is published through no fault of the PI or Institution, or was in the possession of the PI or Institution at time of disclosure and was not acquired from Sponsor under any obligation of confidentiality or is produced pursuant to a validly issued subpoena.